CLINICAL TRIAL: NCT06712862
Title: A Clinical Study of Evaluating Myocardial Viability in Ischemic Heart Disease with Integrated 18F-FDG PET/MR
Status: Recruiting | Type: Observational
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022097
Record Dates: First submitted 2024-11-27; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Ischemic Heart Disease
Keywords: PET/CMR; Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Research group: All patients will receive an integrated 18F-FDG PET/MR scan within 2 weeks before surgery.
- Control Group: All patients will receive integrated 18F-FDG PET/MR plus 99mTc MIBI G-MPI (gated myocardial perfusion imaging) within 2 weeks before surgery.

SUMMARY:
The main purpose is to evaluate the accuracy of myocardial imaging obtained through integrated 18F-FDG PET/MR in detecting viable myocardium. The secondary objective is to evaluate whether myocardial imaging obtained through integrated 18F-FDG PET/MR can replace 18F-FDG PET combined with 99mTc MIBI SPECT/CT gated myocardial perfusion imaging.

DETAILED DESCRIPTION:
A comprehensive evaluation of the degree of coronary artery stenosis, myocardial ischemia range, and survival status are required before surgery, which can help predict postoperative efficacy and select the best treatment plan. Only when the heart muscle is alive, can the myocardial blood flow return to normal after revascularization surgery, improving left ventricular ejection fraction (LVEF) and long-term survival rate of patients. Performing coronary artery bypass grafting(CABG) on patients with lack of myocardial activity not only cannot benefit them, but also increases the risk of surgery. At present, the combination of 18F-flurodeoxyglucose(FDG) Positron Emission Tomography/ Computed Tomography(PET/CT) imaging and myocardial perfusion imaging is the most commonly used method in clinical practice to determine myocardial activity based on the matching of metabolism and blood flow. In recent years, the value of Cardiovascular Magnetic Resonance(CMR) in ischemic diagnosis and myocardial infarction assessment has been widely clinically validated, and many techniques in CMR have been included in clinical guidelines. Late Gadolinium Enhancement(LGE) imaging is the most accurate non-invasive technique for evaluating myocardial scars currently. Integrated Positron Emission Tomography/Magnetic Resonance imaging(PET/MR) can simultaneously evaluate myocardial perfusion, metabolism, vitality, and function, which has certain value for the diagnosis of myocardial ischemia and clinical prognosis of revascularization surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adults under the age of 80
2. Coronary angiography shows coronary artery disease, with at least 2 coronary arteries having a degree of stenosis greater than 80%
3. ft ventricular ejection fraction (LVEF)<40%
4. Acute myocardial infarction onset for at least 3 months
5. Patients with old myocardial infarction with no acute coronary artery events in the past 3 months
6. Patients of pre implementation of coronary artery bypass grafting (CABG) or combined treatment with human umbilical cord mesenchymal stem cells (iPSC)
7. Agree to participate in this clinical trial and sign an informed consent form
8. Good compliance

Exclusion Criteria:

* 1.Patients with diabetes or other patients with poor blood glucose control (fasting blood glucose value on the test day is greater than 10mmol/L) 2.Patients who allergy to MR contrast agent 3.Electronic implants such as pacemakers, nerve stimulators, insulin pumps, cochlear implants 4.Patients who have undergone aneurysm surgery and have intracranial aneurysm clips 5.Patients who have undergone heart surgery and have an artificial heart valve 6.Patients with metal foreign objects in the eyes 7.Patients with metal implants and prostheses, or metal foreign bodies in other parts of body 8.Severe liver and kidney dysfunction 9.Accompanied by arrhythmia such as atrial fibrillation, cerebrovascular disease, and severe pulmonary heart disease 10.Pregnant or plan to pregnant within three months or lactating women 11.Critically ill patients who require the use of life support systems 12.Patients with claustrophobia 13.Other situations which clinical trial personnel deem it inappropriate to participate in this trial

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who meet the inclusion and exclusion criteria and are willing to follow the research process.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Myocardial perfusion tomographic imaging | After the patient signs the informed consent form and completes the scan, an average of 2 days.
  In accordance with the guidelines established by the American Heart Association, the left ventricular myocardium is segmented into 17 distinct regions and subjected to visual assessment for the identification of reversible myocardial perfusion abnormalities or defects.
Myocardiac metabolic Imaging | After the patient signs the informed consent form and completes the scan, an average of 2 days.
  In accordance with the guidelines established by the American Heart Association, the left ventricular myocardium is partitioned into 17 segments, which are subsequently assessed for the presence of diminished myocardial FDG uptake.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
To protect patient privacy, we will not share data. But if the researcher has reasonable reasons, they can apply to the research leader via email.